CLINICAL TRIAL: NCT01725490
Title: The Chemopreventive Effect of Metformin in Patients With Familial Adenomatous Polyposis: Double Blinded Randomized Controlled Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4-2012-0491
Record Dates: First submitted 2012-10-31; First posted 2012-11-12 (Estimated); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Familial Adenomatous Polyposis
Keywords: chemoprevention, metformin, familial adenomatous polyposis
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- metformin 500mg daily (arm A) (Experimental)
  Interventions: Drug: Metformin
- metformin 1500mg daily (arm B) (Experimental)
  Interventions: Drug: Metformin
- an identical- appearing placebo (arm C) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Patients will be randomly assigned in a 2:2:1 ratio to receive metformin or identical-appearing placebo tablets orally for 7 months: metformin 500mg once and placebo twice a day in arm A, metformin 500mg three times a day in arm B, and placebo three times a day in arm C.
  Arms: metformin 500mg daily (arm A)
Drug: Metformin — Patients will be randomly assigned in a 2:2:1 ratio to receive metformin or identical-appearing placebo tablets orally for 7 months: metformin 500mg once and placebo twice a day in arm A, metformin 500mg three times a day in arm B, and placebo three times a day in arm C.
  Arms: metformin 1500mg daily (arm B)
Drug: Placebo — Patients will be randomly assigned in a 2:2:1 ratio to receive metformin or identical-appearing placebo tablets orally for 7 months: metformin 500mg once and placebo twice a day in arm A, metformin 500mg three times a day in arm B, and placebo three times a day in arm C.
  Arms: an identical- appearing placebo (arm C)

SUMMARY:
Familial adenomatous polyposis (FAP) leads to adenomas and eventual adenocarcinomas in colon and less frequently, duodenum. Chemopreventive strategies have been studied in FAP patients to delay the development of adenomas and cancers. The non-steroidal anti-inflammatory drugs (NSAIDs) and selective cyclooxygenase-2 inhibitor have shown the regression of colorectal and duodenal adenomas in FAP patients. However, these drugs showed gastrointestinal damage and cardiovascular risks, and new preventive strategies are needed. Metformin, a biguanide, which is widely used for treating diabetes mellitus, has recently been suggested to have a suppressive effect on tumorigenesis via mTOR-inhibiting pathway, and have no significant safety issues in long term use. The investigators devised a double-blind randomized controlled trial to evaluate the effect of metformin on polyps of colorectum and duodenum in non-diabetic FAP patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with familial adenomatous polyposis(FAP) who are 20 to 65 years of age.
2. FAP patients who have colonic or duodenal polyp
3. FAP patients who have five or more polyps 2mm or more in diameter in endoscopic examination.

Exclusion Criteria:

1. FAP patients who had a history of colectomy within the previous 12 months or need to undergo colectomy within 8 months after randomization.
2. FAP patients with malignant disease, including colorectal cancer.
3. FAP patients who used NSAIDs (non-steroidal anti-inflammatory drugs) or aspirin three or more times a week within 6 months of randomization. 4. FAP patients with diabetes mellitus. 5. Pregnant or breast-feeding patients. 6. Patients with abnormal results of serum laboratory tests (renal function and liver function test) and significant infectious or respiratory diseases.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-02-15 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
the mean percentage change of the number and size of polyps in colon and/or duodenum. | After seven-month administration of metformin/placebo, colonoscopy/sigmoidoscopy and upper gastrointestinal endoscopy will be performed.
  At the base-line endoscopy, India-ink tattoo will be placed in the ascending colon, sigmoid colon/rectum, and duodenum. In case of patient with retained rectum after colectomy and ileorectal anastomosis, sigmoidoscopy will be performed. The base-line and seven-month endoscopic examination will be recorded, and photographs will be taken at the tattoo-marked area and used for measurements of the number and size of polyps. The diameter of a polyp will be measured with the aid of biopsy forceps included in the photographic field, and only distinct polyps at least 2 mm in diameter will be counted.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Park JJ, Kim BC, Hong SP, Seo Y, Lee HS, Park YS, Na SY, Park SC, Park J, Kim JH, Moon CM, Huh KC, Park SJ, Cheon JH, Kim WH, Kim TI. The Effect of Metformin in Treatment of Adenomas in Patients with Familial Adenomatous Polyposis. Cancer Prev Res (Phila). 2021 May;14(5):563-572. doi: 10.1158/1940-6207.CAPR-20-0580. Epub 2021 Jan 28. PMID 33509804